CLINICAL TRIAL: NCT01820676
Title: A Prospective, Multi-Center Study to Evaluate the ConforMIS iUni® G2+ Unicompartmental Knee Resurfacing Device
Brief Title: iUni G2+ Prospective Study
Status: Terminated | Type: Observational
Why Stopped: Decision of investigational team
Sponsor: Restor3D (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-004
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- iUni G2+: iUni G2+ in all patients
  Interventions: Device: iUni G2+

INTERVENTIONS:
Device: iUni G2+ — The iUni G2+ Unicompartmental Resurfacing Device (iUni) is an FDA cleared and CE Marked implant designed for patients with damage isolated to either the medial or lateral tibiofemoral compartment of the knee. The patient-specific iUni is designed from a CT scan of an individual patient's knee using a design process which interactively maps the diseased area and defines the extent of misalignment present in the knee. This process allows definition of the shape and size of the femoral and tibial components of the implant, as well as the disposable instrumentation (Fitz).

SUMMARY:
This study is designed to monitor long term clinical outcomes of the iUni G2+ unicompartmental knee replacement

DETAILED DESCRIPTION:
The study subjects will be followed for 10 years post implant. The follow-up visit schedule will include visits at 6 weeks, 6 months, 1 year, 2 years, 5 years and 10 years post implant.

ELIGIBILITY:
Inclusion Criteria:

* Clinical condition included in the approved Indications For Use
* Unicompartmental osteoarthritis of the medial or lateral tibiofemoral compartment
* Willingness to participate in the clinical study, to give informed consent, and to attend all follow-up visits
* > 18 years of age

Exclusion Criteria:

* Simultaneous bilateral procedure required
* BMI > 35
* Treatment for cancer within the past 5 years, with the exception of skin cancer
* Poorly controlled diabetes
* Neuromuscular conditions which prevent patient from participating in study activities
* Active local or systemic infection
* Immunocompromised
* Fibromyalgia or other general body pain related condition
* Advanced tricompartmental osteoarthritis
* Symptomatic patellofemoral disease
* Rheumatoid arthritis or other forms of inflammatory joint disease (excluding Gout unless it is in the treated knee or limiting overall function)
* Loss of bone or musculature, osteoporosis, osteonecrosis, neuromuscular or vascular compromise in the area of the joint to be operated to an extent that the procedure is unjustified. Osteoporosis is defined by more than -2.5 standard deviations from the T score as measured on a Dual Energy X-Ray Absortiometry Scan (DEXA) within 2 years of surgery.
* Advanced loss of osteochondral structure on the affected femoral condyle
* Compromised ACL, PCL or collateral ligament
* Severe (>15º) fixed valgus or varus deformity
* Extension deficit > 15 º
* Prior history of failed implant surgery of the joint to be treated
* Unwilling or unable to comply with study requirements
* Participation in another clinical study which would confound results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2013-07-15 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
2011 Knee Society Score | 1 Year
KOOS Score | 1 Year
Oxford Knee Score | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Nathwani, MD, Principal Investigator — The London Clinic
Locations (1):
- The London Clinic, London, United Kingdom